CLINICAL TRIAL: NCT06109480
Title: Effect of High Definition Transcranial Direct Current Stimulation (HD-tDCS) Assisted Electroconvulsive Therapy (ECT) for Depression Disorder
Brief Title: Effect of HD-tDCS Assisted ECT for Depression Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-ECT-TDCS-MDD
Record Dates: First submitted 2023-10-21; First posted 2023-10-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Transcranial Direct Current Stimulation; Electroconvulsive Therapy; Depressive Disorder
Keywords: Transcranial Direct Current Stimulation; Electroconvulsive therapy; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ECT combined with real stimulation tDCS group (Active Comparator): Bifrontal short-pulse ECT was performed once a day for 3 consecutive days. Then,tDCS stimulates the dorsomedial prefrontal cortex. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. 2-mA (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes Twice a day over 10 consecutive sessions.
  Interventions: Device: High definition transcranial direct current stimulation; Device: electroconvulsive therapy device
- ECT combined with sham stimulation tDCS group (Sham Comparator): Bifrontal short-pulse ECT was performed once a day for 3 consecutive days. Then,Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: Sham High definition transcranial direct current stimulation; Device: electroconvulsive therapy device
- ECT full course group (Other): The ECT full corse group was used as a standard control.Bifrontal short-pulse ECT was performed once a day for 3 consecutive days,and then once every other day, for a total of 6 times.
  Interventions: Device: electroconvulsive therapy device

INTERVENTIONS:
Device: High definition transcranial direct current stimulation — tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, constant current applied directly to the head through scalp electrodes.
  Arms: ECT combined with real stimulation tDCS group
Device: Sham High definition transcranial direct current stimulation — Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: ECT combined with sham stimulation tDCS group
Device: electroconvulsive therapy device — ECT induces brief generalized epileptic seizures by electric current to stimulate the forehead under general anesthesia

SUMMARY:
To investigate the intervention effect of high definition transcranial direct current stimulation (HD-tDCS) assisted Electroconvulsive Therapy (ECT) for depressive disorder.

DETAILED DESCRIPTION:
Depression is a mental disorder characterized by low mood, decreased interest, and reduced activity. It affects approximately 350 million people around the world and has become a major public health and social problem. Electroconvulsive therapy (ECT) can quickly and effectively improve depressive symptoms, but it causes severe impairment of cognitive functions, such as reduced face memory. Therefore, improving treatment options is of great significance.

Electroconvulsive therapy depends on the number of treatments, usually 2-3 times a week, for a total of 6-12 treatments. Studies have shown early mood improvement after the third ECT. The investigators propose a new ECT treatment strategy, which involves sequential hybridization of high definition transcranial direct current stimulation (HD-tDCS) after the third ECT to maintain its efficacy while mitigating cognitive side effects.

60 patients with depressive disorder diagnosed by Diagnostic and Statistical Manual of Mental Disorders(DSM-5) were recruited from the fourth people's Hospital of Hefei and the Second Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before treatments. After meeting the inclusion criteria and obtaining informed consent, All the participants were randomized (1:1:1) into three groups: ECT combined with real stimulation tDCS group, ECT combined with sham stimulation tDCS group, and ECT full course group.

For ECT combined with real stimulation tDCS group, Bifrontal short-pulse ECT was performed once a day for 3 consecutive days. Then,tDCS stimulates the dorsomedial prefrontal cortex. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. 2 milliampere(mA) (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes Twice a day over 10 consecutive sessions.

For ECT combined with sham stimulation tDCS group,Bifrontal short-pulse ECT was performed once a day for 3 consecutive days.Then,Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.

For ECT full course group,Bifrontal short-pulse ECT was performed once a day for 3 consecutive days, then once every other day, for a total of 6 times,as a traditional contrast Emotional and memory function assessments were conducted at three time points: baseline, post-ECT, and post-TDCS. Emotional assessments included Hamilton Rating Scale for Depression(HAMD), Hamilton Anxiety Scale(HAMA), Beck Scale For Suicide Ideation(BSS), Patient Health Questionnaire-15(PHQ15), Ruminative Responses Scale(RRS), The Temporal Experience of Pleasure Scale (TEPS) and The Positive and Negative Affect Scale(PANAS). Memory function assessments included association memory and working memory.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for depression, and HAMD>17.
* Meets the ECT treatment indication
* the age ranged from 18 to 60 years old, and the length of education was more than 5 years.
* the visual acuity or corrected visual acuity is normal, right-handed, can cooperate with the completion of various experimental tests.

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.
* accompanied by other neurological diseases, such as stroke, epilepsy and so on. pregnant and lactating women.
* accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective disorder, hysteria, autism and so on.
* with a history of ECT treatment within the past 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD) Score | baseline, the third day(immediately after the ECT intervention),the eighth day(immediately after the tDCS intervention)
  The HAMD is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
Change in Associative Memory | baseline, the third day(immediately after the ECT intervention),the eighth day(immediately after the tDCS intervention)
  The associative memory was estimated using a face-cued word association test. In the face-cued word association test, participants studied 12 human face photographs presented individually in grayscale on a computer screen for 4 s per face. Each photograph displayed a unique common word that the participants read aloud as each face-word pair was shown. The participants were instructed to memorize the word associated with each face. After the face-word pairs were presented, participants were shown the same 12 faces, individually and in a different and randomized order. They were asked to recall the words that were presented with each face. Each face was scored as correct or incorrect.These processes are carried out 2 times in total.The average number of successful answers was defined as the associative memory score.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Scale (HAMA) Score | baseline, the third day(immediately after the ECT intervention),the eighth day(immediately after the tDCS intervention)
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
Change in the Patient Health Questionnaire-15 (PHQ-15) scale | baseline, the third day(immediately after the ECT intervention),the eighth day(immediately after the tDCS intervention)
  The PHQ-15 is a 15-item scale to measure the severity of somatic symptoms, where each item is rated on a scale from 0 to 2. The PHQ-15 total score ranges from 0 to 30, with lower scores indicating less somatic symptoms.
Change in Working Memory | baseline, the third day(immediately after the ECT intervention),the eighth day(immediately after the tDCS intervention)
  The n-back task is one of the most common tasks in working memory studies, involving the storage and manipulation of information. In the 2-back condition, they were required to press a button when the current stimulus matched the stimulus from two trials back; in the 1-back condition, participants pressed a button if the current stimulus matched the immediately preceding stimulus.The n-back task consisted of two block-design functional runs, each of which lasted 336 s.Each run included four block sets, where the 1-back and 2-back conditions were intermixed. The order of blocks in each run was pseudorandomized across participants.The average correct rate in the two conditions was used as an indicator of working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghua Tian, PhD, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, China